CLINICAL TRIAL: NCT04876859
Title: Conventional Radiofrequency of Anterior Sensory Branches in Chronic Hip Pain Due to Hip Osteoarthritis: A Randomized Clinical Trial
Brief Title: Comparative Study Between Steroid Plus Anesthetic Block and CRF in Participants With Hip Osteoarthritis
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Main researcher changed institutions, making it unfeasible to be completed by the others participants.
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, João Luiz Q. Durigan, Professor, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE: 40347320.1.1001.0025
Record Dates: First submitted 2021-04-26; First posted 2021-05-07 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Hip Osteoarthritis; Chronic Pain
MeSH Terms: conditions — Osteoarthritis, Hip; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Radiofrequency Group (Active Comparator): Will be submitted to an anesthetic block of the sensory branches of femoral and obturator nerves to the hip, with 1 ml of 1% lidocaine with 1ml of steroid (Betamethasone Dipropionate 5 mg/ml + Betamethasone Sodium Phosphate 2 mg/ml) for each branch, followed by denervation with CRF (22¬gauge 5¬mm active tip cannula, 10cm in length) with the tip temperature set at 90° C in a single cycle of 90 min.
  Interventions: Procedure: CRF of anterior sensitive branches to the hip
- Anesthetic plus steroid group (Sham Comparator): The sham group will be submitted to the same anesthetic block as described in the intervention group, followed by a simulation of CRF use.
  Interventions: Procedure: Anesthetic block with steroid injection of anterior sensitive branches to the hip

INTERVENTIONS:
Procedure: CRF of anterior sensitive branches to the hip — Steroid and anesthetic extra articular injection followed by denervation using CRF at 90 celsius degree during a period 90 minutes at the sensitive branches of obturator and femoral nerve, separately.
  Arms: Conventional Radiofrequency Group
Procedure: Anesthetic block with steroid injection of anterior sensitive branches to the hip — Corticosteroid and anesthetic extra articular injection at the sensitive branches of obturator and femoral nerve, only
  Arms: Anesthetic plus steroid group

SUMMARY:
This will be a prospective, multi-center, double-blinded, randomized study designed to compare the efficacy of Conventional Radiofrequency (CRF) and the anesthetic block of the anterior sensory branches to the hip to control pain and improve function related to hip osteoarthritis.

DETAILED DESCRIPTION:
This prospective, double-blinded (participant and outcome assessor) clinical trial was designed to investigate the results of the intervention Continuous Radiofrequency (CRF) in the treatment of participants with chronic hip pain secondary to hip osteoarthritis. Participants will be randomized in a 2-arm, parallel groups. The intervention group will be submitted to an anesthetic block of the sensory branches of femoral and obturator nerves to the hip, with 1 ml of 1% lidocaine with 1ml of steroid (Betamethasone Dipropionate 5 mg/ml + Betamethasone Sodium Phosphate 2 mg/ml) for each branch, followed by denervation with CRF (22¬gauge 5¬mm active tip cannula, 10cm in length) with the tip temperature set at 90° C in a single cycle of 90 min. The sham group will be submitted to the same anesthetic block, followed by a simulation of CRF use. The surgeon performing the procedures will only be informed of the randomization after completing the anesthetic block on the participants to avoid bias at its accuracy. Participants will be evaluated at four follow-up: before intervention and after 1, 12, and 24 weeks, to access the Western Ontario and McMaster Universities score (WOMAC) as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years or older
* Symptomatic unilateral hip osteoarthritis (OA)
* Pain for more than 6 months in the groin, anterior, anterolateral ou lateral region
* OA radiologically classified as Kellgren and Lawrence Tipo II-IV,
* VAS ≥ 4
* Considered non-responder to conservative treatment for the participant for 6 months.
* In case of difficulty in selecting participants with symptomatic unilateral OA, symptomatic bilateral hip OA will be admitted and submitted to the same treatment on both sides, after notification and approval from the Ethic Board of each institution involved.

Exclusion Criteria:

* Participants with radiculopathy ipsolateral
* Knee OA ipsolateral,
* Previous hip arthroplasty
* Pain exclusively in the posterior region of the hip
* Infiltration of the hip for less than 3 months
* Neurological disease compromising gait
* Peripheral neuropathy
* Psychiatric disease that compromise collaboration with the protocol
* Implanted pacemaker
* Prothrombin Activity Time (PT/INR) > 3 and
* Litigation process related to the disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (WOMAC) | Baseline to 24 weeks ± 1 week.
  The Western Ontario and McMaster Universities (WOMAC) is a self-administered health status measure and consists of 24 items divided into three domains, which are pain (5 questions), stiffness (2 questions), and physical function (17 questions), validated to patients with hip or knee osteoarthritis, available in a 5-point Likert scale, ranging from 0 to 96 points.This questionnaire is translated and validated in portuguese.

SECONDARY OUTCOMES:
Change in Pain Visual Analogue Scale | Baseline, 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  The pain visual analogue scale (VAS) is a unidimensional measure of pain intensity, in a continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme, "no pain" (score 0) and " worst pain ever" (score 100).
Change in Harris Hip Score (HHS) | Baseline, 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  The Harris Hip Score (HHS) is a joint-specific measure, and it consists of two sections: questions and a physical examination, including a range of motion and deformity items. The score has a maximum of 100 points with a maximum of 44 points for pain, 47 for function, 4 points for absence of deformity, and 5 points for a range of motion. The highest score of 100 points indicates the best function and no pain.
Pain Medication Intake | Baseline, 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  To evaluate pain medication we will use a scale ranging from 0 to 4 (0= no medication; 0 = no medication; 1= use of dipyrone or paracetamol; 2= use of NSAIDs; 3= use of opiate derivatives; 4= routinely scheduled opiate derivatives), considering the last 48 hours.
Change in Hip muscles Isometric Peak Force | Baseline, 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  To examine isometric muscle force, a Lafayette Manual Muscle Testing System Model-01165 (Lafayette Instrument Company, Lafayette IN, USA) will be used to access Peak Force of hip flexors, abductors, adductors and extensors.
Change in Hip muscles Time to Reach Peak Force | Baseline, 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  To examine isometric muscle force, a Lafayette Manual Muscle Testing System Model-01165 (Lafayette Instrument Company, Lafayette IN, USA) will be used to access Time to Reach Peak Force of hip flexors, abductors, adductors and extensors.
Change in Hip muscles Average Force | Baseline, 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  To examine isometric muscle force, a Lafayette Manual Muscle Testing System Model-01165 (Lafayette Instrument Company, Lafayette IN, USA) will be used to access Average Force of hip flexors, abductors, adductors and extensors. We will also determine intra and inter-rater reliability for isometric force of hip flexors, abductors, adductors and extensors.
Evaluation of intra and inter-rater reliability of Lafayette Manual Muscle Testing System Model-01165 in subjects with hip Osteoarthritis. | Baseline
  To determine intra and inter-rater reliability of the Hand lend dynamometer Lafayette Manual Muscle Testing System Model-01165 (Lafayette Instrument Company, Lafayette IN, USA) in accessing peak force, time to reach peak force and average force of hip flexors, abductors, adductors and extensors, the first 20 participants included in this study will be evaluated by the principal investigator and outcome assessor at the baseline.
Change in Global Satisfaction | 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  To evaluate participant satisfaction, we will use 5 points Likert Scale, ranging from 0 to 4 (0= none _ no good at all, ineffective intervention; 1= poor _ some effect but unsatisfactory; 2= fair _ reasonable effect but could be better; 3= good _ satisfactory effect with occasional episodes of pain or stiffness; 4= excellent _ ideal response, virtually pain-free).

OTHER OUTCOMES:
Incidence of Adverse Effects | 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  To examine the incidence of adverse effects, a questionnaire will be apply to investigate the occurrence of: Hematoma, paresthesia, weakness, worsening of pain, worsening of function or any other adverse effect that participants attribute to the procedure performed.

CONTACTS AND LOCATIONS:
Overall Officials: João Durigan, PhD, Study Director — Universidade de Brasilia
Locations (1):
- Hospital das Forças Armadas, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Undecided